CLINICAL TRIAL: NCT06734481
Title: Effectiveness and Safety of Sodium Bicarbonate Pleural Lavage in the Treatment of Complex Pleural Effusion: Protocol for a Multicenter Randomized Controlled Trial（SAPLIC Study）
Brief Title: Effectiveness and Safety of Sodium Bicarbonate Pleural Lavage in the Treatment of Complex Pleural Effusion
Acronym: SAPLIC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital of Ningbo University (Network)
Responsible Party: Principal Investigator, Caochao, Principal Investigator, First Affiliated Hospital of Ningbo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-R006-01
Record Dates: First submitted 2024-12-09; First posted 2024-12-16 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Complicated Pleural Effusion/ Empyema

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Saline group (Placebo Comparator): Participants will receive a daily intrapleural injection of 200 mL of saline in 7 days besides standard antibiotic therapy.
  Interventions: Drug: Saline pleural lavage
- Sodium bicarbonate group (Experimental): Participants will receive a daily intrapleural injection of 200 mL of 2.5% sodium bicarbonate in 7 days besides standard antibiotic therapy.
  Interventions: Drug: Sodium bicarbonate pleural lavage

INTERVENTIONS:
Drug: Sodium bicarbonate pleural lavage — All participants will receive a standardized antimicrobial therapy regimen, with antibiotics selected based on susceptibility testing. Within 2 days of initiating treatment, all patients will undergo catheter placement for continuous drainage of pleural effusion. Participants will receive a daily intrapleural injection of 200 mL of 2.5% sodium bicarbonate in 7 days. For patients with ultrasound evidence of pleural effusion loculations or drainage tube obstruction, intrapleural administration of urokinase may be performed at the discretion of the treating physician to ensure effective drainage.Following each daily injection, the catheter will be clamped for 2 hours before resuming continuous drainage, a process that will continue for 7 days.
  Arms: Sodium bicarbonate group
Drug: Saline pleural lavage — All participants will receive a standardized antimicrobial therapy regimen, with antibiotics selected based on susceptibility testing. Within 2 days of initiating treatment, all patients will undergo catheter placement for continuous drainage of pleural effusion. Participants will receive a daily intrapleural injection of 200 mL of saline in 7days For patients with ultrasound evidence of pleural effusion loculations or drainage tube obstruction, intrapleural administration of urokinase may be performed at the discretion of the treating physician to ensure effective drainage. Following each daily injection, the catheter will be clamped for 2 hours before resuming continuous drainage, a process that will continue for 7 days..
  Arms: Saline group

SUMMARY:
The goal of this clinical trial is to evaluate the safety and efficacy of sodium bicarbonate pleural lavage in treating complex pleural effusion in adult. The main questions it aims to answer are:

Will sodium bicarbonate pleural lavage reduce the failure rate of medical treatment (referral rate for surgery) for complicated pleural effusion？ Can sodium bicarbonate pleural lavage accelerating the rehabilitation of patients with complicated pleural effusion？ Will sodium bicarbonate pleural lavage improve the prognosis of patients with complicated pleural effusion?

Participants will will undergo catheter placement for continuous drainage of pleural effusion. Once at least 200 mL of pleural effusion has been drained:

Group A: Participants will receive a daily intrapleural injection of 200 mL of saline in 7 days; Group B: Participants will receive a daily intrapleural injection of 200 mL of 2.5% sodium bicarbonate in 7 days.

DETAILED DESCRIPTION:
For patients with ultrasound evidence of pleural effusion loculations or drainage tube obstruction, intrapleural administration of urokinase may be performed at the discretion of the treating physician to ensure effective drainage.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients aged 18 to 80 years, inclusive.
* Patients fulfilling any one of the following three criteria for complicated pleural effusion: A. Pleural fluid pH < 7.2; B. Pleural fluid glucose < 2.2 mmol/L and LDH > 1000 IU/L; C. Positive pleural fluid culture or smear for pathogens.
* Pleural effusion volume exceeding 300 mL, as determined by CT imaging using the formula D^2 * L (where D represents the maximum depth and L the maximum length), and for whom pleural effusion drainage is clinically indicated according to established guidelines or criteria.

Exclusion Criteria:

* Patients with known allergies to sodium bicarbonate or normal saline.
* Patients with severe coagulation disorders.
* Patients with severe heart or kidney failure.
* Pregnant or lactating women.
* Patients with pleural effusion caused by hospital-acquired interference, tuberculosis, fungal infections, or non-infectious causes.
* Patients unable to tolerate intrapleural administration.
* Patients with chronic lung diseases that may affect antibiotic efficacy, such as uncontrolled chronic obstructive pulmonary disease (COPD GOLD E group), bronchiectasis, or immunodeficiency.
* Patients who have experienced shock, major bleeding, trauma, or pulmonary surgery within the past 5 days.
* Patients with a history of lung or pleural surgery on the side of the pleural effusion.
* Patients who have recently had chest tubes placed due to pneumothorax, surgery, or pleural effusion.
* Patients currently enrolled in another drug or device clinical trial.
* Patients with poor compliance or difficulty in follow-up, or those with an expected survival of less than 3 months due to conditions other than pleural effusion.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Failure rate of medical treatment (referral rate for surgery) | Week 2.

SECONDARY OUTCOMES:
Change in Pleural Thickness Before and After Treatment | Baseline, week 2, week 12 and 3-month follow up.
Volume of Pleural Effusion Before and After Treatment | Baseline, week 2, week 12 and 3-month follow up.
Average Length of Hospital Stay | Up to 3 months.
Inflammatory Response at 1 Week and 2 Weeks Post-Treatment | Baseline, week 1 and week 2.
All-Cause Mortality | Up to 3 months.

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affiliated Hospital of Ningbo University, Ningbo, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No